CLINICAL TRIAL: NCT04697082
Title: Application of Platelet-rich Plasma for the Management of Pilonidal Sinus Disease: A Randomized Clinical Trial of Different Treatment Modalities
Brief Title: Application of Platelet-rich Plasma in Pilonidal Sinus Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cihangir Akyol (Other)
Responsible Party: Sponsor-Investigator, Cihangir Akyol, Associate Proffessor, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1263-3749
Record Dates: First submitted 2021-01-01; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Pilonidal Sinus; Pilonidal Disease; Wound Heal; Quality of Life; Pain
Keywords: PRP; Wound healing; Pilonidal sinus; Quality of life; Pain
MeSH Terms: conditions — Pilonidal Sinus; Pain | interventions — Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: The patients were divided into three groups randomly. A simple randomization diagram was used for randomization.
  The open surgical method and a moist dressing were applied to patients in group A.
  Open surgery and then PRP application were performed on patients in group B. PRP was applied to the patients in group C after curettage of the sinus cavity.
  49 patients were included in the analysis. In this study, we compared the impact of autologous platelet-rich plasma (PRP) with that of minimally invasive techniques on pain reduction, return to daily activities, quality of life, and duration of wound healing after open excision and secondary closure.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): The open surgical method and a moist gauze (with saline) were applied to patients in group A
  Interventions: Procedure: Open surgery
- Group B (Experimental): Open surgery and then PRP application were performed on patients in group B. After the cavity was filled with PRP, the wound was covered with a dry gauze.
  Interventions: Procedure: Open surgery; Other: Platelet rich plasma administration
- Group C (Experimental): PRP was applied to the patients in group C after curettage of the sinus cavity. And again the wound was covered with a dry gauze.
  Interventions: Procedure: Minimal invasive surgery; Other: Platelet rich plasma administration

INTERVENTIONS:
Procedure: Open surgery — Each patient entered the operating room, and after the administration of general anaesthesia, the patient was placed in the prone position. Then, the buttocks were stretched to the lateral sides using adhesive bands to remove the disease area. The sacrococcygeal region was cleaned and disinfected with 10% povidone iodine. After covering the area around the region, the sinus tract was examined by using a thin-steel cane. The length and wealth of the cavity were noted. Then, the sinus tract was removed. The depth of the cavity was noted. Then, 50 cc of 0.9% saline solution (SS) was taken into a syringe and applied to the cavity until it filled the whole space, allowing the cavity volume to be measured accurately. The measurement was performed by subtracting the remaining saline-solution volume in the syringe from the whole syringe volume, which was 50 cc.
  Arms: Group A; Group B
Procedure: Minimal invasive surgery — In the operating room, after the patient was placed in the prone position, the region was removed by stretching the buttocks with adhesive bands and cleaning the area with 10% povidone iodine. The largest pit was excised, and hairs in the cavity were removed with forceps. Then, the whole cavity was curetted meticulously and irrigated with SS. After haemostasis, the cavity volume was measured
  Arms: Group C
Other: Platelet rich plasma administration — Platelet rich plasma (PRP) was administered by filling the whole space from the lateral side of the cavity. After the first implementation of PRP, the second one was applied at 48 hours. Until that time, the dressing was not uncovered. PRP was applied on the 3rd, 4th and 5th days postoperatively.
  Arms: Group B; Group C

SUMMARY:
Pilonidal sinus disease is a common health-care problem, and surgical excision is the standard treatment modality. Controversy still exists regarding the best surgical technique for treating pilonidal disease in terms of minimizing disease recurrence and patient discomfort. In this study, the investigators compared the impact of autologous platelet-rich plasma (PRP) with that of minimally invasive techniques on pain reduction, return to daily activities, quality of life, and duration of wound healing after open excision and secondary closure.

DETAILED DESCRIPTION:
Pilonidal sinus disease is a health problem that has been attempted to be overcome by various treatment modalities since the first time it was described by Herbert Mayo in 1833. PS is usually diagnosed at 30 years of age, and the disease has a male predominance of 70-80%.

Common morbidities after the surgical treatment of PS are pain, loss of productive work hours and wound infections owing to long healing times. Therefore, the main goals of treatment are accelerating the healing time by decreasing pain and reducing the loss of productive work hours.

Local administration of platelet-rich plasma (PRP), which contains growth factors (Gfs), is a new method that has been reported to accelerate the healing process by 30-40% [2].

In this study, we aimed to investigate the effect of PRP on the pain score, wound-healing process and quality of life in the treatment process for PS disease.

METHOD

Trial Design The investigators designed the trial as a prospective, controlled-randomized study. The study was started after obtaining patient consent and approval from the Ethics Committee of Ankara University Medicine Faculty in Ankara (Ethics Committee no: 03-162-18).

Randomization The patients were divided into three groups randomly. A simple randomization diagram was used for randomization. The open surgical method and a moist dressing were applied to patients in group A. Open surgery and then PRP application were performed on patients in group B. PRP was applied to the patients in group C after curettage of the sinus cavity.

Medical and Demographic History After enrolling the patients, the investigators noted all demographic data, including gender, age, education, comorbid disease existence and drug use. Then, Short Form-36 (SF-36) and Nottingham Health Profile (NHP) quality-of-life score forms were given to the patients, who were asked to complete the questionnaires before the surgery.

All patients were asked to clean the sacrococcygeal region from hair using depilatory cream.

Surgical Procedure The investigators designed group A as the control group. In this group, each patient entered the operating room, and after the administration of general anaesthesia, the patient was placed in the prone position. Then, the buttocks were stretched to the lateral sides using adhesive bands to remove the disease area. The sacrococcygeal region was cleaned and disinfected with 10% povidone iodine. After covering the area around the region, the sinus tract was examined by using a thin-steel cane. The length and wealth of the cavity were noted. Then, the sinus tract was removed. The depth of the cavity was noted. Then, 50 cc of 0.9% saline solution (SS) was taken into a syringe and applied to the cavity until it filled the whole space, allowing the cavity volume to be measured accurately. The measurement was performed by subtracting the remaining saline-solution volume in the syringe from the whole syringe volume, which was 50 cc. After measurement of the cavity volume, the cavity was dressed with wet gauze, and the operation ended.

PRP Administration Group B was designed as local PRP administration after excision. Whole steps were applied the same as in the first group until the step of dressing the cavity. After measurement of the cavity volume with 0.9% SS, PRP was administered by filling the whole space from the lateral side of the cavity. After the first implementation of PRP, the second one was applied at 48 hours. Until that time, the dressing was not uncovered. PRP was applied on the 3rd, 4th and 5th days postoperatively.

Minimal Invasive Surgery Group C was designed to receive local PRP administration after minimally invasive surgery with local anaesthesia. In the operating room, after the patient was placed in the prone position, the region was removed by stretching the buttocks with adhesive bands and cleaning the area with 10% povidone iodine. The largest pit was excised, and hairs in the cavity were removed with forceps. Then, the whole cavity was curetted meticulously and irrigated with SS. After haemostasis, the cavity volume was measured, and PRP was applied to the cavity. After the first implementation, as in the second group, we applied PRP on the 2nd, 3rd, 4th and 5th days after surgery.

Preparation of PRP For clinical applications, GMP-compliant human platelet concentrates can be created by the PRP method. Erythrocyte concentrate and platelet-containing plasma are separated by the first centrifugation, and platelet-poor plasma (PPP) and platelet-rich plasma (PRP)/platelet concentrate are created by the second centrifugation of the platelet-containing plasma [3]. Platelets contain coagulation factors, growth factors (PDGF, TGFβ1, IGF1, HGF1, VEGF, FGF2) and interleukins (IL1, IL4, IL6, IL10, IL13) [4].

The investigators prepared the platelet concentrate by the PRP method in Hacettepe University Blood Center Laboratory considering all standardized processes for healthy blood donors. In accordance with the 'National Blood and Blood Components Preparation Use and Quality Assurance Guidelines', the requirements for PRP should include at least 40 mL in volume, at least 60x109/unit platelets [5], and a maximum of 0.2x109/unit leukocytes [6]. After approval, 450 cc of blood was drawn from the patient by phlebotomy on the morning of surgery. A two-stage centrifugation method was used in the process of separating complete blood into its components. In the first stage, plasma was separated with the erythrocyte suspension by using temperature-controlled Heraeus Cryofuge 6000i low-speed centrifugation (22°C, 2500 rpm, 7 minutes). After a 1-hour waiting period at the second stage, the PRP/platelet concentrate was separated from the PPP by using high-speed centrifugation (22°C, 3200 rpm, 15 minutes). The PRP/platelet concentrate obtained after the second centrifugation step was shaken in the agitator for 1 hour, divided into 5 equal parts with a sterile connection device (Figure) and then sent to the Ankara University General Surgery Department.

The investigators preserved the PRP at 25 degrees Celsius in agitators. Before each dressing, the investigators applied the PRP aliquots to the wound by taking them one by one into the injector.

Postoperative Care All patients were discharged on the first postoperative day. Patients in all groups were advised not to open the wound for 2 days. Additionally, the surgical area had to be kept clean after bathing and bowel movements. If the patients experienced pain, they were recommended to take the prescribed pain reliever no more than 2 times a day.

ELIGIBILITY:
Inclusion Criteria:

* chronic pilonial sinus disease
* patients who had undergone abscess drainage and remained diseased after 8-10 weeks of drainage

Exclusion Criteria:

* patients with acute abscess
* patients with anemia
* patients that use immunosuppressive drugs
* patients with haematological malignancy
* patients with bleeding disorder
* patients with recurrent pilonida sinus disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Wound Healing | on postoperative days 0, 2, 3, 4 and 21
  Wound healing rate was evaluated as recovery time per the cavity volume (day/cc). This showed the time required for each 1 cc volume of the cavity to be filled on a daily basis. After open or minimally invasive surgery, the volume of the cavity was measured with saline solution. The cavity was filled with saline and the volume of the cavity was determined by calculating how much fluid it took. The measurements were performed on postoperative days 0, 2, 3, 4 and 21. Therefore recovery time per the cavity volume was calculated according to the differences between the measurements.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) score | at 24th hour, 48th hour, 96th hour, 120th hour and 3rd week
  We used a visual analogue scale (VAS) to evaluate the pain score. The VAS score can range from 0 to 10. The higher the score, the higher sensation of pain. The VAS was applied five times after surgery: at 24 hours, 48 hours, 96 hours, 120 hours and 3 weeks. Patients were routinely prescribed "dexketoprofen trometamol" and recommended to take it no more than 2 times a day. How many tablets the patients used after the operation was recorded.
Short Form-36 and Nottingham Health Profile | before the surgery and in the postoperative 3rd week
  Short Form-36 (SF-36) and Nottingham Health Profile (NHP) questionnaires were applied to evaluate the quality of life before the surgery and three weeks after.
  The SF-36 consists of eight scaled scoresand each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
  The NHP consists of two parts. The highest score in any section is 100 The higher the score, the greater the number and severity of problems We assessed the general health, limitations or activities, physical health problems, emotional health problems, social activity, pain, energy and emotions of the patients with the SF-36 questionnaire. Additionally, we evaluated the pain, energy level, emotional reaction, sleep, social isolation, and physical abilities of patients with the NHP questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Can Y Boztug, MD, Principal Investigator — Ankara University School of Medicine Departmernt of General Surgery; Cihangir Akyol, MD, Study Chair — Ankara University School of Medicine Departmernt of General Surgery
Locations (1):
- Ankara University School of Medicine Department of General Surgery, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boztug CY, Karaagac Akyol T, Benlice C, Koc MA, Doganay Erdogan B, Ozcebe OI, Kuzu MA, Akyol C. Platelet-rich plasma treatment improves postoperative recovery in patients with pilonidal sinus disease: a randomized controlled clinical trial. BMC Surg. 2021 Oct 21;21(1):373. doi: 10.1186/s12893-021-01370-5. PMID 34670534